CLINICAL TRIAL: NCT02373683
Title: Helium-oxygen Gas Mixtures Delivered by a High Flow Nasal Cannula in Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Katherine Slain, DO, Case Western Reserve University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-14-08
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Bronchiolitis; Heliox; Pediatrics
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapotherm-Heliox (Experimental): Following separation from mechanical ventilation, patient is placed on heliox (70% oxygen-30% helium) delivered with Vapotherm, a proprietary heated, humidified, high-flow nasal cannula delivery system.
  Interventions: Device: Vapotherm-Heliox
- Standard Care (No Intervention): Care dictated by clinical team.

INTERVENTIONS:
Device: Vapotherm-Heliox — Following separation from mechanical ventilation, patient is placed on heliox (70% oxygen-30% helium) delivered with Vapotherm, a proprietary heated, humidified, high-flow nasal cannula delivery system.
  Arms: Vapotherm-Heliox

SUMMARY:
The aim of this prospective pilot study is to determine the effect of heliox delivered via a proprietary calibrated heated and humidified high flow nasal cannula (HFNC) system (Vapotherm Precision Flow Heliox) in children ages 0-24 months with severe bronchiolitis.

DETAILED DESCRIPTION:
Respiratory syncytial virus associated bronchiolitis is a leading cause of global infant morbidity and mortality [1], yet care remains largely supportive. Several recent studies show that a helium-oxygen gas mixture (heliox) improves outcomes in children with moderate to severe bronchiolitis [2-5, 7]. Heliox is a safe, inert gas with no biological effects and very low density [6]. By improving laminar flow, heliox improves gas exchange in conditions where airway resistance is increased, such as asthma, croup and bronchiolitis [6].

Recent data shows that infants with moderate to severe bronchiolitis have a reduced length of hospital stay when heliox is delivered via facemask or CPAP, as compared to heliox via nasal cannula [2]. Limitations to this study include the small number of patients (84/319 [26%]) who tolerated the facemask therapy and the fact that nasal cannula heliox was delivered at low flows (3 LPM). Oxygen is increasingly being delivered with a heated, humidified, high flow nasal cannula (HFNC) system to infants with moderate to severe bronchiolitis in our PICU. To date, there are no definitive randomized controlled trials that show the HFNC system is an effective treatment in bronchiolitis. However, there are several retrospective, prospective and pilot interventional studies showing clinical improvement in this patient population treated with the HFNC system [8-11]. We hypothesize that delivering heliox via a heated, humidified, high flow nasal cannula will be well tolerated, safe and effective.

Specific Aim #1: The aim of this prospective pilot study is to determine the effect of heliox delivered via a proprietary calibrated heated and humidified high flow nasal cannula (HFNC) system (Vapotherm Precision Flow Heliox) in children ages 0-24 months with severe bronchiolitis.

Hypothesis #1: Clinical and physiologic markers of respiratory distress will be improved in patients receiving heliox via HFNC compared to standard therapy following separation from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-24 months
* Admission to the Pediatric Intensive Care Unit
* Diagnosis of bronchiolitis, with respiratory syncytial virus infection confirmed by laboratory testing
* Mechanical ventilation

Exclusion Criteria:

* Inclusion in another clinical trial
* Significant cardiac disease
* Anatomically abnormal airway
* Neurologic disease
* Immunodeficiency
* History of chronic lung disease
* Craniofacial anomaly
* Chromosomal anomalies
* Known or suspected dysphagia

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Rotta, MD, Principal Investigator — Rainbow Babies and Children's Hospital, University Hospitals Case Medical Center
Locations (1):
- Rainbow Babies Children's Hospital, University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Background] Chowdhury MM, McKenzie SA, Pearson CC, Carr S, Pao C, Shah AR, Reus E, Eliahoo J, Gordon F, Bland H, Habibi P. Heliox therapy in bronchiolitis: phase III multicenter double-blind randomized controlled trial. Pediatrics. 2013 Apr;131(4):661-9. doi: 10.1542/peds.2012-1317. Epub 2013 Mar 18. PMID 23509160
- [Background] Martinon-Torres F, Rodriguez-Nunez A, Martinon-Sanchez JM. Heliox therapy in infants with acute bronchiolitis. Pediatrics. 2002 Jan;109(1):68-73. doi: 10.1542/peds.109.1.68. PMID 11773543
- [Background] Kim IK, Phrampus E, Sikes K, Pendleton J, Saville A, Corcoran T, Gracely E, Venkataraman S. Helium-oxygen therapy for infants with bronchiolitis: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Dec;165(12):1115-22. doi: 10.1001/archpediatrics.2011.605. PMID 22147778
- [Background] Gupta VK, Cheifetz IM. Heliox administration in the pediatric intensive care unit: an evidence-based review. Pediatr Crit Care Med. 2005 Mar;6(2):204-11. doi: 10.1097/01.PCC.0000154946.62733.94. PMID 15730610
- [Background] Liet JM, Ducruet T, Gupta V, Cambonie G. Heliox inhalation therapy for bronchiolitis in infants. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD006915. doi: 10.1002/14651858.CD006915.pub2. PMID 20393951
- [Background] Abboud PA, Roth PJ, Skiles CL, Stolfi A, Rowin ME. Predictors of failure in infants with viral bronchiolitis treated with high-flow, high-humidity nasal cannula therapy*. Pediatr Crit Care Med. 2012 Nov;13(6):e343-9. doi: 10.1097/PCC.0b013e31825b546f. PMID 22805160
- [Background] Bressan S, Balzani M, Krauss B, Pettenazzo A, Zanconato S, Baraldi E. High-flow nasal cannula oxygen for bronchiolitis in a pediatric ward: a pilot study. Eur J Pediatr. 2013 Dec;172(12):1649-56. doi: 10.1007/s00431-013-2094-4. Epub 2013 Jul 31. PMID 23900520
- [Background] Milesi C, Baleine J, Matecki S, Durand S, Combes C, Novais AR, Cambonie G. Is treatment with a high flow nasal cannula effective in acute viral bronchiolitis? A physiologic study. Intensive Care Med. 2013 Jun;39(6):1088-94. doi: 10.1007/s00134-013-2879-y. Epub 2013 Mar 14. PMID 23494016
- [Background] Schibler A, Pham TM, Dunster KR, Foster K, Barlow A, Gibbons K, Hough JL. Reduced intubation rates for infants after introduction of high-flow nasal prong oxygen delivery. Intensive Care Med. 2011 May;37(5):847-52. doi: 10.1007/s00134-011-2177-5. Epub 2011 Mar 3. PMID 21369809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vapotherm-Heliox | Standard Care
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was not collected or analyzed for enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vapotherm-Heliox | Standard Care | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: months] — Population: Data was not collected or analyzed.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data was not collected or analyzed
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary diagnosis [Count of Participants; unit: Participants] — Population: Data was not collected or analyzed

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Assessment Score
Description: Change in the respiratory assessment score from baseline (within 15 minutes of extubation) to 48 hours after extubation. The score ranges from 0 to 12, with higher scores indicating worsening respiratory distress.
Time Frame: 48 hours
Population: Study was terminated early. Data were not collected and results were not analyzed.
Arm/Group | Vapotherm-Heliox | Standard Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Need for Reintubation
Time Frame: During hospitalization, typically 4 days to 2 weeks
Population: Study was terminated early. Data were not collected and results were not analyzed.
Arm/Group | Vapotherm-Heliox | Standard Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: PICU Length of Stay
Time Frame: During hospitalization, typically 4 days to 2 weeks
Population: Study was terminated early. Data were not collected and results were not analyzed.
Arm/Group | Vapotherm-Heliox | Standard Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Time Frame: During hospitalization, typically 4 days to 2 weeks
Population: Study was terminated early. Data were not collected and results were not analyzed.
Arm/Group | Vapotherm-Heliox | Standard Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Length of Treatment With Supplemental Oxygen
Time Frame: During hospitalization, typically 4 days to 2 weeks
Population: Study was terminated early. Data were not collected and results were not analyzed.
Arm/Group | Vapotherm-Heliox | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vapotherm-Heliox | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes